CLINICAL TRIAL: NCT01681966
Title: A Single-dose, Open-Label, Multi-center Study to Assess the Safety and Preliminary Efficacy of PRF 110 (Formerly LNP) in Open Herniorrhaphy Surgery
Brief Title: A Single-dose Open-Label Study to Assess the Safety and Preliminary Efficacy of PRF 110 in Open Herniorrhaphy Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PainReform LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNP-IL102
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Application of PRF110- oily solution (Experimental): Post operative application of new extended release PRF110- oily solution (Ropivacaine)
  Interventions: Drug: PRF110- oily solution (Ropivacaine)

INTERVENTIONS:
Drug: PRF110- oily solution (Ropivacaine) — Post operative application of PRF110-oily solution (Ropivacaine)
  Other Names: Ropivacaine oily solution

SUMMARY:
LNP is new extended release (ER) oily solution formulation of ropivacaine that is intended for local infiltration into surgical wounds. The purpose of this study is to determine the ease of usage and administration of LNP in the surgical setting, to follow the Pharmacokinetic (PK) profile of LNP over 72 hours and evaluate the duration of analgesia witnessed in the surgical setting.

DETAILED DESCRIPTION:
LNP is new extended release (ER) oily solution formulation of ropivacaine that is intended for local infiltration into surgical wounds. The formulation is designed to slowly release the ropivacaine over 36-72 hours. By providing local analgesia over a long time span, the need for systemic analgesics is expected to be reduced and hospital stays may be shortened. The purpose of this study is to determine the ease of usage and administration of LNP in the surgical setting, to follow the PK profile of LNP over 72 hours and evaluate the duration of analgesia witnessed in the surgical setting.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between 18-70 years of age who are scheduled to undergo open one sided herniorrhaphy surgery;
* Subjects have a BMI of less than 30 kg/m2;
* Subjects are in good physical health (other than the need for the surgical procedure) as judged by physical and laboratory examinations and have a negative urine based screen for drugs of abuse;
* Subjects must agree to refrain from ingesting any analgesic medication for at least 2 days (or 5 half-lives of the analgesic drug) prior to surgery; refrain from alcohol and excessive caffeine intake on the day of surgery and during 72 hours after surgery;
* Subject must be capable of reading, comprehending, and signing the informed consent form;

Exclusion Criteria:

* Subjects with a history of melena or any significant hepatic, renal, endocrine, cardiac, neurological, psychiatric, gastrointestinal, pulmonary, hematologic, or metabolic disorders;
* Subjects with a history of any type of cancer within 5 years of surgery;
* Subjects with any history of alcohol or substance abuse;
* Subjects that have a history of uncontrolled hypertension;
* Subjects with a known hypersensitivity to any local anesthetic drug;
* Subjects with a hemoglobin concentration of less than 10.0 g/dL;
* Subjects with any clinically significant abnormal lab result (as judged by the Principal Investigator);
* Subjects with atrial fibrillation/flutter, an inserted pacemaker, or complete left bundle branch block (LBBB) on ECG; or myocardial infarction within 6 months prior to surgery;
* Subjects with a clinically significant abnormal ECG at screening;
* Subjects with any condition or history judged by the Investigator to place the subject at increased risk;
* Subjects judged by the Investigator to be unable or unwilling to comply with the requirements of the protocol;
* Subjects who have used an investigational drug within 30 days prior to entering the study;
* Subjects who have donated blood within 3 months prior to the start of the study;
* Subjects who are members of the study site staff directly involved with the study or a relative of the Sponsor or other personnel involved with the study;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09; Primary Completion 2016-05-04 (Actual); Study Completion 2016-05-04 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (safety and tolerability). | 72 hours
  All adverse events (AE) reported by the subjects will be recorded throughout the trial period

SECONDARY OUTCOMES:
Post-operative Pain intensity | 72 hours
  Pain on a scale of 0-10 assessed at 0,1,2,4,8,12,24,36,48,60,72hrs post operation will be used to evaluate pain intensity

OTHER OUTCOMES:
Use of rescue medication | 72 hours
  Overall use of rescue medication post operation
Maximum plasma concentration (Cmax) | 72 hrs
  Samples will be collected at designated times up to 72hrs post drug application

CONTACTS AND LOCATIONS:
Overall Officials: Moaad Farraj, Dr., Principal Investigator — Galilee Medical Center
Locations (3):
- Israel (3):
  - Western Galil Medical Center, Nahariya
  - Assaf Harofeh Medical Center, Rishon LeZiyyon
  - Sourasky Medical Center, Tel Aviv